CLINICAL TRIAL: NCT06054191
Title: A Phase II, Two Parallel Group Study of Neoadjuvant and Adjuvant Targeted Treatment in NSCLC With BRAF V600 or MET Exon 14 Mutations
Brief Title: Neoadjuvant and Adjuvant Targeted Treatment in NSCLC With BRAF V600 or MET Exon 14 Mutations
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, MD, Director, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2023-331-01
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: NSCLC; BRAF V600 Mutation; MET Exon 14 Mutation
MeSH Terms: interventions — dabrafenib; trametinib; capmatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: BRAF V600 mutation (Experimental): Dabrafenib + Trametinib
  Interventions: Drug: Dabrafenib + Trametinib
- Cohort 2: MET ex14 skip mutation (Experimental): Capmatinib
  Interventions: Drug: Capmatinib

INTERVENTIONS:
Drug: Dabrafenib + Trametinib — Dabrafenib 150mg BID + Trametinib 2mg QD/（2 cycles）
  Arms: Cohort 1: BRAF V600 mutation
Drug: Capmatinib — Capmatinib 400mg BID/（2 cycles）
  Arms: Cohort 2: MET ex14 skip mutation

SUMMARY:
This is a Phase II, two parallel group study assessing the efficacy and safety of neoadjuvant and adjuvant targeted therapy in patients with stage IB-IIIA NSCLC harboring BRAF V600 or MET exon14 mutations.

DETAILED DESCRIPTION:
This is a Phase II, two parallel group study assessing the efficacy and safety of neoadjuvant and adjuvant targeted therapy in patients with stage IB-IIIA NSCLC harboring BRAF V600 or MET exon14 mutations. Eligible patients with BRAF V600 mutations will receive dabrafenib 150mg bid plus trametinib 2mg qd for 8 weeks before a surgical resection (neoadjuvant), and followed by up to 4 cycles of adjuvant chemotherapy, if receive adjuvant chemotherapy, up to four cycles, chemo regimen according to investigators' choice, and up to 2 years of adjuvant targeted therapy with dabrafenib plus trametinib. For patients with MET exon14 mutations, they will receive capmatinib 400mg bid for 8 weeks before surgery (neoadjuvant), followed by up to 4 cycles of adjuvant chemotherapy, about adjuvant chemotherapy same as BRAF V600 group, and up to 2 years of adjuvant targeted therapy with capmatinib post-surgery. During treatment, patients will visit their physicians regularly for disease and safety assessment. After the end of treatment, survival follow-up will be conducted every 3 months for up to 3 years. Approximately 40 evaluable patients will be enrolled in the study (20 patients in each cohort).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Histologically or cytologically diagnosed stage IB-IIIA and selected IIIB (T3N2, T4N2) NSCLC.
* Presence of BRAF V600 mutation or METex14 skip mutation in tumor (by PCR or NGS) or blood (by NGS) (pre-treatment biopsy confirmed) in local or other Clinical Laboratory Improvement Amendments (CLIA)-certified lab.
* Patients whose pre-surgical lesion is measurable, Eligible for surgical resection and scheduled for surgery within 2 weeks after the last does of neoadjuvant treatment.
* ECOG performance-status score of 0 or 1.
* No previous anticancer therapy.
* Patients with stage II or higher non-small-cell lung cancer (NSCLC) and those with suspected brain metastases should have brain imaging (CT or MRI) prior to enrollment to exclude brain metastasis.
* Could provide pretreatment tumor samples available for biomarker analysis. The subject should have good compliance, who would participate in the research voluntarily, and sign the informed consent.

Exclusion Criteria:

* Patients with unresectable (regardless of stage) or metastatic disease (stage IV) or brain metastases.
* Contain neuroendocrine carcinoma tumor histology.
* Major surgery within 4 weeks before enrollment, or who have not recovered from side effects of related procedures.
* History of current interstitial lung disease or pneumonitis.
* Patients with conditions requiring systemic corticosteroids (>10 mg daily prednisone or equivalent) or immunosuppressive medication within 14 days of the first dose of study drug (Inhaled or topical steroids and adrenal-replacement steroids are allowed).
* History of other malignancies within 5 years (excluding basal cell carcinoma of the skin or other carcinoma in situ that has been resected).
* Pregnant or lactating women.
* Those who are allergic to the research drug or its components.
* Subjects who are deemed unable to comply with the study requirements or complete the study.
* Those with acquired immunodeficiency syndrome, or any uncontrolled medical disorder, or insufficient function of bone marrow or other important organs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | up to 2 years
  pCR rate is defined as the percentage of participants with no residual viable tumor cells.

SECONDARY OUTCOMES:
Major pathological response (MPR) rate | up to 2 years
  MPR rate is defined as the percentage of participants with ≤10% residual viable tumor cells.
Event-free survival (EFS) | up to 3 years
  EFS is defined as the time from intervention to the first documented disease progression per RECIST v1.1 that precludes surgery, local or distant disease recurrence, or death from any cause, whichever occurs first.
Disease-free survival (DFS) | up to 3 years
  DFS defined as the time from the end of surgery until recurrence or death due to any cause, DFS rate at 12, 24, 36 and 60 months.
Overall survival (OS) | up to 3 years
  OS defined as the time between the date of enrollment and the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center of Sun-Yat Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided